CLINICAL TRIAL: NCT02202317
Title: Follow-up Yttrium-90 Internal Pair Production PET/CT Imaging in Patients With Primary or Metastatic Liver Tumors as Compared With Brehmsstrahlung Imaging: A Prospective Case Series
Brief Title: Follow-up Yttrium-90 Internal Pair Production PET/CT vs Brehmsstrahlung Imaging in Patients With Primary/Metastatic Liver Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jason Salsamendi, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20120092
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Results first posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Liver Cancer; Hepatic Tumors
Keywords: Liver Cancer; Hepatic Tumors; Primary Liver Tumors; Metastatic Liver Tumors; Yttrium-90; Y-90
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Positron Emission Tomography Computed Tomography

ARMS (1):
- Y90 Based PET/CT Scan (Experimental)
  Interventions: Device: PET/CT Scan

INTERVENTIONS:
Device: PET/CT Scan — Subjects will receive a PET/CT Scan in addition to SPECT imaging, from the level of the lower chest to the lower pelvis, typical of an abdominal CT, usually within 1-3 hours after Yttrium-90 treatment.

SUMMARY:
This is a prospective non-blinded case series involving the acquisition of a pair production PET/CT as soon as possible after an already performed Y-90 Sirspheres treatment of hepatic malignancy. It will be performed in addition to the standard Brehmsstrahlung SPECT scan. The sequence of the two scans in each case (PET/CT vs SPECT) will be determined by availability of the scanners at the time. However, it is intended that both be acquired on the day of the Y-90 treatment.

The length of subject participation will be one year.

The measures used will be mostly qualitative in nature, and will include:

* Correlation with expected vs. achieved tumor coverage by the treatment
* Correlation between treatment distribution depicted by Brehmsstrahlung scans vs. the Internal Pair Production PET/CT scans, to.
* Detection of non-target embolization, where applicable, and qualitative comparison between the two modalities as to the conspicuity of the abnormality

Qualitative methods will be used by the analysis of the obtained PET/CT images and comparing them to the Brehmsstrahlung SPECT images as previously described.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of Selective Internal Radiation Treatment within 5 days.
* Anticipated ability to remain still for up to 40 minutes

Exclusion Criteria:

* Anticipated Inability to lie still for up to 40 minutes
* Severe claustrophobia
* Significant cardiovascular instability, or instability of other medical/surgical conditions, such that it would be deemed unsafe or technically not feasible to obtain a PET/CT, as determined by the any member of the investigative team
* Failed deployment of the planned Y-90 treatment for any reason
* Duration of time longer than 5 days since administration of the Y-90 treatment
* Age <18
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Salsamendi, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Health System, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Y90 Based PET/CT Scan
Started | 9
Completed | 8
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The initial number of patients that participated in the study is 9. However, one patient elected not to return for the PET/CT scan after Y-90 delivery, therefore the total number of participants analyzed is 8 patients.
Arm/Group | Y90 Based PET/CT Scan
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Whose Y-90 Based PET/CT (Positron Emission Tomography/Computed Tomography)Scans Detected Extrahepatic Non-target Embolization.
Description: Number of participants with detected extrahepatic non-target embolization. A qualitative comparison between the two modalities (Y-90 PET/CT and Brehmsstrahlung SPECT) as to the conspicuity of the abnormality would have been conducted had any participant had that result.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Y90 Based PET/CT Scan
Number analyzed (Participants) | 8
Participants | 0

2. Secondary Outcome: Comparison Between Treatment Distribution Depicted by Tc99mMAA (Technetium-99m Macroaggregated Albumin) Brehmsstrahlung Scans vs. the Internal Pair Production PET/CT Scans.
Description: Number of participants demonstrating a similar treatment distribution depicted by Tc99mMAA(Technetium-99m macroaggregated albumin) Brehmsstrahlung scans vs. achieved Y-90 distribution on the Internal Pair Production PET/CT scans.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Y90 Based PET/CT Scan
Number analyzed (Participants) | 8
Participants | 8

3. Secondary Outcome: Comparison of Y-90 PET/CT to Y90 SPECT
Description: Number of participants with a similar Y90 distribution depicted on Post Y90 delivery PET/CT and SPECT modalities, specifically comparing Y90 distribution within the treated tumors.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Y90 Based PET/CT Scan
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Arm/Group | Y90 Based PET/CT Scan
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No